CLINICAL TRIAL: NCT00497146
Title: The PRIMO Study: Paricalcitol Capsules Benefits in Renal Failure Induced Cardiac Morbidity in Subjects With Chronic Kidney Disease Stage 3/4
Brief Title: The PRIMO Study: Paricalcitol Capsules Benefits Renal Failure Induced Cardiac Morbidity in Subjects With Chronic Kidney Disease Stage 3/4
Acronym: PRIMO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M10-030; 2007-001689-34 (EudraCT Number)
Record Dates: First submitted 2007-07-03; First posted 2007-07-06 (Estimated); Results first posted 2011-12-23 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Chronic Kidney Disease; Left Ventricular Hypertrophy
Keywords: paricalcitol; Zemplar; PRIMO; Chronic Kidney Disease Stage 3B/4
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertrophy, Left Ventricular | interventions — paricalcitol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paricalcitol (Experimental): Participants received paricalcitol capsules 2 µg once a day (two 1 µg paricalcitol capsules), for up to 48 weeks. Participants who completed the 48-week Treatment Period could continue in the Long-term Follow-up Period for an additional 18 months. Participants did not receive study drug during the Long-term Follow-up Period.
  Interventions: Drug: paricalcitol
- Placebo (Placebo Comparator): Participants received 2 placebo capsules once a day for up to 48 weeks. Participants who completed the 48-week Treatment Period could continue in the Long-term Follow-up Period for an additional 18 months. Participants did not receive study drug during the Long-term Follow-up Period.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: paricalcitol — 2 µg capsule
  Other Names: ABT-358; Zemplar
  Arms: Paricalcitol
Drug: placebo — placebo capsule
  Arms: Placebo

SUMMARY:
To evaluate the effects of paricalcitol capsules on cardiac structure and function over 48 weeks in patients with Stage 3/4 chronic kidney disease (CKD) who had left ventricular hypertrophy (LVH).

DETAILED DESCRIPTION:
Patients who met the inclusion criteria and did not meet any of the exclusion criteria were randomized in a 1:1 ratio to each treatment group to receive paricalcitol capsules or placebo. A stratified randomization scheme was used to ensure balance among treatment groups with respect to country, gender, and baseline renin angiotensin-aldosterone system (RAAS) inhibitor use (yes/no).

Participants who completed the 48-Week Treatment Period could continue on in the ongoing Long-term Follow-up Period that was to last 18 months, with study visits at 6 months, 12 months and 18 months post Treatment Week 48 Visit. Participants did not receive study drug, nor were they to have undergone echocardiogram/MRI procedures during the Long-term Follow-up Period.

ELIGIBILITY:
Inclusion Criteria:

* Estimated glomerular filtration rate (GFR) between 15-60 mL/min/1.73 m^2
* Serum intact parathyroid hormone (iPTH) value between 50-300 pg/mL
* Corrected serum calcium level 8.0-10.0 mg/dL (2.0-2.5 mmol/L)
* Phosphorous level less than or equal to 5.2 mg/dL (1.68 mmol/L)
* Serum albumin greater than or equal to 3.0 g/dL (30 g/L)
* Echocardiogram results of:

  * Females: Left ventricular (LV) ejection fraction greater than or equal to 50% and septal wall thickness between 11-17 mm; and,
  * Males: LV ejection fraction greater than or equal to 50% and septal wall thickness between 12-18 mm
* If the subject is receiving renin-angiotensin-aldosterone system (RAAS) inhibitors the dose must have been stable for greater than one month prior to the Screening Period. However, the subject may have switched to different brands but at equivalent doses as determined by the study physician during the month prior to the Screening Period.
* Subject must have a technically adequate baseline cardiac magnetic resonance imaging (MRI).

Exclusion Criteria:

* Subject has previously been on active vitamin D therapy within the four weeks prior to the Screening Period
* Pregnant or lactating females
* Subject is expected to initiate renal replacement therapy within one year
* Subject is taking calcitonin, bisphosphonates, cinacalcet, glucocorticoids (except topical or inhaled glucocorticoids)
* Subject had clinically significant coronary artery disease (CAD) within 3 months prior to the Screening Period, defined as either hospitalization for myocardial infarction (MI) or unstable angina; new onset angina with positive functional study or coronary angiogram revealing stenosis; or coronary revascularization procedure.
* Subject had major cardiac valve abnormality linked with LVH and/or diastolic dysfunction, defined as either aortic valve area ≤ 1.5 cm^2 or a mean gradient of > 20 mmHg; or regurgitation lesions; more than moderate mitral regurgitation, or more than moderate aortic regurgitation.
* Subject had asymmetric septal hypertrophy defined as septal wall thickness/posterior wall thickness ratio > 1.5 based on screening echocardiogram.
* Subject had a severe cerebrovascular accident (CVA) within the last 3 months (e.g., hemorrhagic) prior to screening.
* Subject had full remission from a malignancy for less than 1 year except completely excised non-melanoma skin cancer (e.g., basal or squamous carcinoma) or any history of bone metastasis.
* Subject had comorbid conditions (e.g., advanced malignancy, advanced liver disease) with a life expectancy less than 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2008-02; Primary Completion 2010-09 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Eldred, MD, Study Director — AbbVie
Locations (71):
- United States (30):
  - Site Reference ID/Investigator# 8062, Phoenix, Arizona
  - Site Reference ID/Investigator# 8867, Tempe, Arizona
  - Site Reference ID/Investigator# 8864, San Diego, California
  - Site Reference ID/Investigator# 7257, San Dimas, California
  - Site Reference ID/Investigator# 7727, Denver, Colorado
  - Site Reference ID/Investigator# 8861, Miami, Florida
  - Site Reference ID/Investigator# 7260, Orlando, Florida
  - Site Reference ID/Investigator# 7725, Tampa, Florida
  - Site Reference ID/Investigator# 7824, Tampa, Florida
  - Site Reference ID/Investigator# 18882, Meridian, Idaho
  - Site Reference ID/Investigator# 7823, Chicago, Illinois
  - Site Reference ID/Investigator# 7249, Evergreen Park, Illinois
  - Site Reference ID/Investigator# 7816, Bethesda, Maryland
  - Site Reference ID/Investigator# 18881, Rockville, Maryland
  - Site Reference ID/Investigator# 7817, Springfield, Massachusetts
  - Site Reference ID/Investigator# 7245, Detroit, Michigan
  - Site Reference ID/Investigator# 7248, Royal Oak, Michigan
  - Site Reference ID/Investigator# 8868, Kansas City, Missouri
  - Site Reference ID/Investigator# 7828, St Louis, Missouri
  - Site Reference ID/Investigator# 14442, Omaha, Nebraska
  - Site Reference ID/Investigator# 6567, Winston-Salem, North Carolina
  - Site Reference ID/Investigator# 7262, Winston-Salem, North Carolina
  - Site Reference ID/Investigator# 7826, Allentown, Pennsylvania
  - Site Reference ID/Investigator# 8865, Chattanooga, Tennessee
  - Site Reference ID/Investigator# 7261, Houston, Texas
  - Site Reference ID/Investigator# 8058, Houston, Texas
  - Site Reference ID/Investigator# 7830, San Antonio, Texas
  - Site Reference ID/Investigator# 7825, Murray, Utah
  - Site Reference ID/Investigator# 8866, Provo, Utah
  - Site Reference ID/Investigator# 7263, Fairfax, Virginia
- Australia (6):
  - Site Reference ID/Investigator# 8493, Adelaide
  - Site Reference ID/Investigator# 8506, Liverpool
  - Site Reference ID/Investigator# 8507, Parkville
  - Site Reference ID/Investigator# 9581, Reservoir
  - Site Reference ID/Investigator# 9582, Richmond
  - Site Reference ID/Investigator# 8500, Westmead
- Czechia (3):
  - Site Reference ID/Investigator# 8245, Prague
  - Site Reference ID/Investigator# 8246, Prague
  - Site Reference ID/Investigator# 8499, Prague
- Germany (5):
  - Site Reference ID/Investigator# 6692, Dortmund
  - Site Reference ID/Investigator# 9723, Düsseldorf
  - Site Reference ID/Investigator# 6630, Lübeck
  - Site Reference ID/Investigator# 7268, Nettetal
  - Site Reference ID/Investigator# 6622, Würzburg
- Italy (3):
  - Site Reference ID/Investigator# 10626, Lido di Camaiore
  - Site Reference ID/Investigator# 8070, Naples
  - Site Reference ID/Investigator# 8060, Rome
- Site Reference ID/Investigator# 8519, Lodz, Poland
- Puerto Rico (6):
  - Site Reference ID/Investigator# 7702, Humacao
  - Site Reference ID/Investigator# 7269, Ponce
  - Site Reference ID/Investigator# 7818, Rio Piedras
  - Site Reference ID/Investigator# 7270, San Juan
  - Site Reference ID/Investigator# 7712, San Juan
  - Site Reference ID/Investigator# 7266, Toa Baja
- Romania (3):
  - Site Reference ID/Investigator# 8881, Bucharest
  - Site Reference ID/Investigator# 8518, Bucharest
  - Site Reference ID/Investigator# 8514, Iași
- Russia (4):
  - Site Reference ID/Investigator# 22682, Moscow
  - Site Reference ID/Investigator# 8009, Moscow
  - Site Reference ID/Investigator# 7251, Moscow
  - Site Reference ID/Investigator# 7250, Moscow
- Spain (5):
  - Site Reference ID/Investigator# 8883, Barcelona
  - Site Reference ID/Investigator# 8358, Barcelona
  - Site Reference ID/Investigator# 8355, Madrid
  - Site Reference ID/Investigator# 8356, Madrid
  - Site Reference ID/Investigator# 8882, Santander (Cantabria)
- Taiwan (4):
  - Site Reference ID/Investigator# 8884, Taipei
  - Site Reference ID/Investigator# 8228, Taipei
  - Site Reference ID/Investigator# 8229, Taoyuan District
  - Site Reference ID/Investigator# 8234, Xinzhuang
- Site Reference ID/Investigator# 8823, Coventry, United Kingdom

REFERENCES:
- [Derived] Tamez H, Zoccali C, Packham D, Wenger J, Bhan I, Appelbaum E, Pritchett Y, Chang Y, Agarwal R, Wanner C, Lloyd-Jones D, Cannata J, Thompson BT, Andress D, Zhang W, Singh B, Zehnder D, Pachika A, Manning WJ, Shah A, Solomon SD, Thadhani R. Vitamin D reduces left atrial volume in patients with left ventricular hypertrophy and chronic kidney disease. Am Heart J. 2012 Dec;164(6):902-9.e2. doi: 10.1016/j.ahj.2012.09.018. Epub 2012 Oct 29. PMID 23194491
- [Derived] Thadhani R, Appelbaum E, Pritchett Y, Chang Y, Wenger J, Tamez H, Bhan I, Agarwal R, Zoccali C, Wanner C, Lloyd-Jones D, Cannata J, Thompson BT, Andress D, Zhang W, Packham D, Singh B, Zehnder D, Shah A, Pachika A, Manning WJ, Solomon SD. Vitamin D therapy and cardiac structure and function in patients with chronic kidney disease: the PRIMO randomized controlled trial. JAMA. 2012 Feb 15;307(7):674-84. doi: 10.1001/jama.2012.120. PMID 22337679
- [Derived] Thadhani R, Appelbaum E, Chang Y, Pritchett Y, Bhan I, Agarwal R, Zoccali C, Wanner C, Lloyd-Jones D, Cannata J, Thompson T, Audhya P, Andress D, Zhang W, Ye J, Packham D, Singh B, Zehnder D, Manning WJ, Pachika A, Solomon SD. Vitamin D receptor activation and left ventricular hypertrophy in advanced kidney disease. Am J Nephrol. 2011;33(2):139-49. doi: 10.1159/000323551. Epub 2011 Jan 18. PMID 21242674
- [Derived] Thadhani R. Targeted ablation of the vitamin D 1alpha-hydroxylase gene: getting to the heart of the matter. Kidney Int. 2008 Jul;74(2):141-3. doi: 10.1038/ki.2008.219. PMID 18591942
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in the study at US and ex-US investigative sites. Recruitment began in March 2008 and ended in December 2009. The study population consisted of participants with Stage 3/4 chronic kidney disease who had a diagnosis of left ventricular hypertrophy confirmed by echocardiogram and cardiac magnetic resonance imaging.
Period: Treatment Period
Arm/Group | Paricalcitol | Placebo
Started | 115 | 112
Completed | 88 | 91
Not Completed | 27 | 21
Not completed — Adverse Event | 6 | 2
Not completed — Withdrawal by Subject | 5 | 9
Not completed — Lost to Follow-up | 1 | 3
Not completed — Required dialysis | 4 | 1
Not completed — Change in RAAS inhibitor therapy | 5 | 2
Not completed — Unable to dose reduce per protocol | 4 | 1
Not completed — Other Reason | 2 | 3
Period: Long-term Follow-up Period
Arm/Group | Paricalcitol | Placebo
Started | 65 | 72
Completed | 50 | 66
Not Completed | 15 | 6
Not completed — Adverse Event | 2 | 2
Not completed — Withdrawal by Subject | 8 | 2
Not completed — Lost to Follow-up | 5 | 1
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paricalcitol | Placebo | Total
Number analyzed (Participants) | 115 | 112 | 227
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 56 | 51 | 107
  >=65 years | 59 | 61 | 120
Age Continuous [Mean (Standard Deviation); unit: years] | 64.3 (11.30) | 65.7 (12.20) | 65.0 (11.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 33 | 69
  Male | 79 | 79 | 158
Baseline RAAS Status [Number; unit: participants] — Baseline renin angiotensin-aldosterone system (RAAS) status refers to whether or not (yes/no) the participant was receiving RAAS inhibitor therapy at baseline.
  participants
    Yes | 90 | 87 | 177
    No | 25 | 25 | 50
Diabetic Status [Number; unit: participants]
  Type I | 4 | 1 | 5
  Type II | 59 | 56 | 115
  None | 52 | 55 | 107
Age at Beginning of Long term Follow-up Period [Mean (Standard Deviation); unit: years] — Age demographics for the long-term follow-up population include data for 65 and 72 participants in the paricalcitol and placebo groups, respectively.
  years | 64.6 (11.01) | 66.5 (12.09) | 65.6 (11.58)
Gender at Beginning of Long term Follow-up Period [Number; unit: participants]
  Female | 20 | 25 | 45
  Male | 45 | 47 | 92

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Left Ventricular Mass Index (LVMI) Over 48 Weeks Measured by Cardiac Magnetic Resonance Imaging (MRI)
Description: The Central Cardiac MRI Core Laboratory (CCL) interpreted and analyzed all cardiac MRI data. Left Ventricular Mass (LVM) was normalized to the participant's height by the following equation to obtain LVMI: LVM (grams) divided by height (meters)^2.7.
Time Frame: Baseline to 48 weeks
Population: The analysis was based on the intent-to-treat (ITT) population, defined as all randomized participants who took at least one dose of study drug, with available data.
Measure: Least Squares Mean (Standard Error); unit: grams/meter^2.7
Arm/Group | Paricalcitol | Placebo
Number analyzed (Participants) | 82 | 87
grams/meter^2.7 | 0.34 (0.248) | -0.07 (0.246)
Statistical Analysis 1: Comparison: Paricalcitol vs Placebo; Test type: Superiority or Other; p = 0.145, Mixed Models Analysis; Mixed model includes treatment, visit, gender, baseline RAAS inhibitor use, country, baseline value, and treatment by visit interaction

2. Secondary Outcome: Change in Diastolic Mitral Annular Relaxation Velocity (E')
Description: Diastolic mitral annular relaxation velocity (lateral E wave velocity; E') is a measure of diastolic function.
Time Frame: Baseline to 48 weeks
Population: The intent-to-treat (ITT) population, participants with available data.
Measure: Least Squares Mean (Standard Error); unit: centimeters/second
Arm/Group | Paricalcitol | Placebo
Number analyzed (Participants) | 79 | 80
centimeters/second | -0.01 (0.314) | -0.30 (0.323)

3. Secondary Outcome: Change in Ratio of Peak E Wave Velocity to Lateral E Wave Velocity (E/E')
Description: The ratio of peak E wave velocity to lateral E wave velocity (E/E') is a measure of diastolic function.
Time Frame: Baseline to 48 weeks
Population: The intent-to-treat (ITT) population, participants with available data.
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Paricalcitol | Placebo
Number analyzed (Participants) | 78 | 77
ratio | 0.16 (0.580) | -0.33 (0.601)

4. Secondary Outcome: Change in E-wave Deceleration Time (DT)
Description: E-wave deceleration time (DT) is a measure of diastolic function.
Time Frame: Baseline to 48 weeks
Population: The intent-to-treat (ITT) population, participants with available data.
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Paricalcitol | Placebo
Number analyzed (Participants) | 82 | 80
seconds | 0.01 (0.004) | -0.00 (0.005)

5. Secondary Outcome: Change in Isovolumetric Relaxation Time (IVRT)
Description: Isovolumetric relaxation time (IVRT) is a measure of diastolic function.
Time Frame: Baseline to 48 weeks
Population: The intent-to-treat (ITT) population, participants with available data.
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Paricalcitol | Placebo
Number analyzed (Participants) | 83 | 81
seconds | 0.00 (0.002) | -0.00 (0.002)

6. Secondary Outcome: Change in Left Atrial Volume
Description: Left atrial volume is a measure of diastolic function.
Time Frame: Baseline to 48 weeks
Population: The intent-to-treat (ITT) population, participants with available data.
Measure: Least Squares Mean (Standard Error); unit: milliliters
Arm/Group | Paricalcitol | Placebo
Number analyzed (Participants) | 82 | 80
milliliters | -4.94 (1.159) | -0.92 (1.193)

7. Secondary Outcome: Change in Plasma Triiodothyronine (T3)
Description: Plasma triiodothyronine (T3) is a biological and inflammatory marker.
Time Frame: Baseline to 48 weeks
Population: The intent-to-treat (ITT) population, participants with available data.
Measure: Least Squares Mean (Standard Error); unit: nanomoles/liter
Arm/Group | Paricalcitol | Placebo
Number analyzed (Participants) | 83 | 87
nanomoles/liter | 0.07 (0.036) | 0.12 (0.036)

8. Secondary Outcome: Change in Interleukin-6 (IL-6)
Description: Interleukin-6 (IL-6) is a biological and inflammatory marker.
Time Frame: Baseline to 48 weeks
Population: The intent-to-treat (ITT) population, participants with available data.
Measure: Least Squares Mean (Standard Error); unit: nanograms/liter
Arm/Group | Paricalcitol | Placebo
Number analyzed (Participants) | 81 | 85
nanograms/liter | 0.27 (0.844) | -0.85 (0.847)

9. Secondary Outcome: Change in Troponin-T
Description: Troponin-T is a biological and inflammatory marker.
Time Frame: Baseline to 48 weeks
Population: The intent-to-treat (ITT) population, participants with available data.
Measure: Least Squares Mean (Standard Error); unit: micrograms/liter
Arm/Group | Paricalcitol | Placebo
Number analyzed (Participants) | 79 | 88
micrograms/liter | 0.01 (0.002) | 0.00 (0.002)

10. Secondary Outcome: Change in B-type Natriuretic Peptide (BNP)
Description: B-type natriuretic peptide (BNP) is a biological and inflammatory marker.
Time Frame: Baseline to 48 weeks
Population: The intent-to-treat (ITT) population, participants with available data.
Measure: Least Squares Mean (Standard Error); unit: log nanograms/liter
Arm/Group | Paricalcitol | Placebo
Number analyzed (Participants) | 79 | 82
log nanograms/liter | 0.19 (0.086) | 0.35 (0.085)

11. Secondary Outcome: Change in High Sensitivity C-reactive Protein (hsCRP)
Description: High sensitivity C-reactive protein (hsCRP) is a biological and inflammatory marker.
Time Frame: Baseline to 48 weeks
Population: The intent-to-treat (ITT) population, participants with available data.
Measure: Least Squares Mean (Standard Error); unit: milligrams/liter
Arm/Group | Paricalcitol | Placebo
Number analyzed (Participants) | 83 | 88
milligrams/liter | 1.49 (1.658) | 1.06 (1.623)

12. Secondary Outcome: Change in Progression of Thoraco-abdominal Aortic Plaque Volume
Description: Change from baseline to Week 48 in thoraco-abdominal aortic plaque volume.
Time Frame: Baseline to 48 weeks
Population: The intent-to-treat (ITT) population, participants with available data.
Measure: Least Squares Mean (Standard Error); unit: milliliters
Arm/Group | Paricalcitol | Placebo
Number analyzed (Participants) | 72 | 72
milliliters | -0.02 (0.002) | -0.03 (0.002)

13. Secondary Outcome: Change in Progression of Thoraco-abdominal Aortic Wall Volume
Description: Change from baseline to Week 48 in thoraco-abdominal aortic wall volume
Time Frame: Baseline to 48 weeks
Population: The intent-to-treat (ITT) population, participants with available data.
Measure: Least Squares Mean (Standard Error); unit: milliliters
Arm/Group | Paricalcitol | Placebo
Number analyzed (Participants) | 75 | 72
milliliters | -0.07 (0.023) | -0.10 (0.024)

14. Secondary Outcome: Change in Progression of Aortic Compliance
Description: Change from baseline to Week 48 in aortic compliance.
Time Frame: Baseline to 48 weeks
Population: The intent-to-treat (ITT) population, participants with available data.
Measure: Least Squares Mean (Standard Error); unit: 10^-4 cm^2/mmHg
Arm/Group | Paricalcitol | Placebo
Number analyzed (Participants) | 78 | 78
10^-4 cm^2/mmHg | -7.24 (5.011) | -5.79 (4.958)

15. Secondary Outcome: Change in Progression of Left Ventricular End-systolic Volume Index
Description: Change from baseline to Week 48 in left ventricular end-systolic volume index.
Time Frame: Baseline to 48 weeks
Population: The intent-to-treat (ITT) population, participants with available data.
Measure: Least Squares Mean (Standard Error); unit: milliliters/meter^2.7
Arm/Group | Paricalcitol | Placebo
Number analyzed (Participants) | 80 | 85
milliliters/meter^2.7 | 0.58 (0.420) | 0.57 (0.412)

16. Secondary Outcome: Change in Progression of Left Ventricular End-diastolic Volume Index
Description: Change from baseline to Week 48 in left ventricular end-diastolic volume index.
Time Frame: Baseline to 48 weeks
Population: The intent-to-treat (ITT) population, participants with available data.
Measure: Least Squares Mean (Standard Error); unit: milliliters/meter^2.7
Arm/Group | Paricalcitol | Placebo
Number analyzed (Participants) | 82 | 87
milliliters/meter^2.7 | 0.30 (0.480) | -0.36 (0.478)

17. Secondary Outcome: Change in Progression of Left Ventricular Ejection Fraction
Description: Change from baseline to Week 48 in left ventricular ejection fraction.
Time Frame: Baseline to 48 weeks
Population: The intent-to-treat (ITT) population, participants with available data.
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Paricalcitol | Placebo
Number analyzed (Participants) | 78 | 79
percent | 0.62 (0.773) | -0.54 (0.771)

ADVERSE EVENTS:
Time Frame: All AE(s) reported from the time of study drug administration until 30 days after last study drug administration were collected (up to 52 weeks). In addition, serious adverse events were collected throughout the 18-month Long-term Follow-up Period.
Description: AEs were coded using the MedDRA version 14.0 coding dictionary for AEs collected during the Treatment Period and version 14.1 for AEs collected during the Long-term Follow-up Period.
Groups:
- Paricalcitol: Treatment Period: Participants received paricalcitol capsules 2 µg once a day (two 1 µg paricalcitol capsules), for up to 48 weeks.
- Placebo: Treatment Period: Participants received 2 placebo capsules once a day for up to 48 weeks.
- Paricalcitol: Long-term Follow-up: Participants who received paricalcitol and completed the 48-week Treatment Period could continue in the Long-term Follow-up Period for an additional 18 months. Participants did not receive study drug during the Long-term Follow-up Period.
- Placebo: Long-term Follow-up: Participants who received placebo and completed the 48-week Treatment Period could continue in the Long-term Follow-up Period for an additional 18 months. Participants did not receive study drug during the Long-term Follow-up Period.
Arm/Group | Paricalcitol: Treatment Period | Placebo: Treatment Period | Paricalcitol: Long-term Follow-up | Placebo: Long-term Follow-up
Serious Adverse Events (participants affected / at risk) | 20/115 | 20/112 | 18/65 | 13/72
Other Adverse Events (participants affected / at risk) | 75/115 | 68/112 | 4/65 | 8/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paricalcitol: Treatment Period (N=115) | Placebo: Treatment Period (N=112) | Paricalcitol: Long-term Follow-up (N=65) | Placebo: Long-term Follow-up (N=72)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 2 | 1 | 2
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 3 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 2 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 3 | 2 | 0
Pneumonia fungal (Infections and infestations) | 1 | 0 | 0 | 0
Scrotal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0
Blood glucose decreased (Investigations) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Diabetic foot (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Nephropathy (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 2 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 2 | 3 | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 1 | 1 | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Aortic dissection (Vascular disorders) | 0 | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0
Autoimmune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1
Aortic valve disease (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Meniere's disease (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Angle closure glaucoma (Eye disorders) | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Small intestine obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Cardiac death (General disorders) | 0 | 0 | 1 | 0
Sudden death (General disorders) | 0 | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Bronchitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1 | 0
Otitis media acute (Infections and infestations) | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Femoral neck injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Tetany (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0
Embolic stroke (Nervous system disorders) | 0 | 0 | 0 | 1
Intracranial haematoma (Nervous system disorders) | 0 | 0 | 1 | 0
Post-traumatic epilepsy (Nervous system disorders) | 0 | 0 | 1 | 0
Azotaemia (Renal and urinary disorders) | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Vesicourteric reflux (Renal and urinary disorders) | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 0 | 0 | 1
Hypertensive emergency (Vascular disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paricalcitol: Treatment Period (N=115) | Placebo: Treatment Period (N=112) | Paricalcitol: Long-term Follow-up (N=65) | Placebo: Long-term Follow-up (N=72)
Anaemia (Blood and lymphatic system disorders) | 7 | 6 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 4 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 3 | 4 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 8 | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 5 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 8 | 5 | 0 | 0
Vomiting (Gastrointestinal disorders) | 4 | 3 | 0 | 0
Asthenia (General disorders) | 3 | 2 | 0 | 0
Chest pain (General disorders) | 3 | 0 | 0 | 0
Fatigue (General disorders) | 6 | 4 | 0 | 0
Oedema peripheral (General disorders) | 2 | 12 | 0 | 1
Bronchitis (Infections and infestations) | 2 | 3 | 0 | 0
Nasopharyngitis (Infections and infestations) | 6 | 7 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 3 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 6 | 5 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 10 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0
Blood creatinine increased (Investigations) | 4 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0
Gout (Metabolism and nutrition disorders) | 4 | 5 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 10 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 4 | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 4 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 5 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 6 | 2 | 0 | 1
Headache (Nervous system disorders) | 5 | 2 | 0 | 0
Lethargy (Nervous system disorders) | 3 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 2 | 3 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 5 | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 4 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 4 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 3 | 0 | 0
Hypertension (Vascular disorders) | 11 | 4 | 0 | 1
Hypotension (Vascular disorders) | 4 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.